CLINICAL TRIAL: NCT00610168
Title: Evaluation of GSK Biologicals' dTpa Booster Vaccine in Young Adults 10 Years After Previous dTpa Boosting.
Brief Title: Immunogenicity & Reactogenicity of Boostrix 10 Years After Previous Booster Vaccination.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110806
Record Dates: First submitted 2008-01-25; First posted 2008-02-07 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2017-02

CONDITIONS: Acellular Pertussis; Tetanus; Diphtheria
Keywords: dTpa vaccine; pertussis; Tdap; Boostrix; booster; tetanus; diphtheria
MeSH Terms: conditions — Tetanus; Diphtheria; Whooping Cough

ARMS (2):
- BOOSTRIX I GROUP (Experimental): Subjects, who had received Boostrix™ vaccine in the primary study (263855/004), received one additional booster dose of Boostrix™ vaccine in this study, administered as an intramuscular injection into the deltoid region of the non-dominant arm.
  Interventions: Biological: Boostrix TM
- BOOSTRIX II GROUP (Experimental): Subjects, who had received Wyeth's (formerly Lederle) combined adult diphtheria and tetanus vaccine and GSK Biologicals' acellular pertussis vaccine in the primary study (263855/004), received one booster dose of Boostrix™ vaccine in this study, administered as an intramuscular injection into the deltoid region of the non-dominant arm.
  Interventions: Biological: Boostrix TM

INTERVENTIONS:
Biological: Boostrix TM — Single booster dose of vaccine
  Other Names: dTpa vaccine

SUMMARY:
The purpose of this study is to assess the efficacy and safety of repeating dTpa booster in adults 10 years after previous booster vaccination with dTpa in a prior clinical study. Only subjects who received booster vaccination in the previous clinical study are eligible for participation in this study.

DETAILED DESCRIPTION:
This Protocol Posting has been updated in order to comply with FDA AA, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* Subjects who have received dTpa vaccine or Td and pa vaccines in study 263855/004.
* A male or female subject, recruited 10 years after booster vaccination in study 263855/004.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential, or, if of childbearing potential, she must use adequate contraception for 30 days prior to vaccination and continue for 2 months after completion of the vaccination series.
* Written informed consent obtained from the subject.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the booster dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the booster dose.
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to booster vaccination or planned administration during the active study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Previous booster vaccination against tetanus, diphtheria or pertussis since the last dose received in study 263855/004.
* History of documented diphtheria, tetanus, or pertussis diseases.
* Any confirmed or suspected immunosuppressive or immunodeficiency condition, based on medical history and physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Administration of immunoglobulins and/or any blood products within the three months preceding the booster dose or planned administration during the study period.
* Occurrence of transient thrombocytopenia or neurological complications following an earlier immunisation against diphtheria and/or tetanus.
* Occurrence of any of the following adverse event after a previous administration of a DTP vaccine :

  * hypersensitivity reaction to any component of the vaccine,
  * encephalopathy of unknown aetiology occurring within 7 days following previous vaccination with pertussis-containing vaccine,
  * fever >= 40°C within 48 hours of vaccination not due to another identifiable cause,
  * collapse or shock-like state (hypotonic-hyporesponsiveness episode) within 48 hours of vaccination,
  * convulsions with or without fever, occurring within 3 days of vaccination.
* Acute disease at the time of enrolment.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions within 2 months after completion of the vaccination series.

Ages: 20 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2008-01-01; Primary Completion 2008-04-30 (Actual); Study Completion 2008-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Turku, Finland

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] He Q et al. Immunity to pertussis 10 years after acellular booster vaccine in adolescence and response to a second dTpa booster in young adults. Abstract presented at the 19th annual european congress of clinical microbiology and infectious diseases, Helsinki, Finland, 16-19 May 2009.
- [Background] Mertsola J, Van Der Meeren O, He Q, Linko-Parvinen A, Ramakrishnan G, Mannermaa L, Soila M, Pulkkinen M, Jacquet JM. Decennial administration of a reduced antigen content diphtheria and tetanus toxoids and acellular pertussis vaccine in young adults. Clin Infect Dis. 2010 Sep 15;51(6):656-62. doi: 10.1086/655825. PMID 20704493
- [Background] Mertsola J et al. Decennial administration of reduced-antigen dTpa vaccine in young adults - incidence of solicited local symptoms classified by pre-vaccination antibody concentrations. Abstract presented at the 27th annual ESPID meeting, Brussels, Belgium, 9-13 June 2009.
- [Background] Mertsola J et al. The immunogenicity and safety of repeated administration of dTpa booster in adolescents and young adults. Abstract presented at the 27th annual ESPID meeting, Brussels, Belgium, 9-13 June 2009.
- [Background] Mertsola J et al. The immunogenicity of repeated administration of reduced-antigen-content dTpa booster in adults. Abstract presented at WSPID-6th World Congress. Buenos Aires, Argentina, 19-22 November 2009
- [Background] Mertsola J et al. The safety of repeated administration of Boostrix™, a reduced-antigen-content dTpa booster. Abstract presented at Excellence In Paediatrics (EIP). Florence, Italy, 3-6 December 2009.
- [Background] Mertsola J et al. The safety of repeated administration of reduced-antigen-content dTpa boosters. Abstract presented at WSPID-6th World Congress. Buenos Aires, Argentina, 19-22 November 2009.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 110806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Boostrix I Group: Subjects, who had received Boostrix vaccine in the primary study (263855/004), received one additional booster dose of Boostrix vaccine in this study, administered as an intramuscular injection into the deltoid region of the non-dominant arm.
- Boostrix II Group: Subjects, who had received Wyeth's (formerly Lederle) combined adult diphtheria and tetanus vaccine and GSK Biologicals' acellular pertussis vaccine in the primary study (263855/004), received one booster dose of Boostrix vaccine in this study, administered as an intramuscular injection into the deltoid region of the non-dominant arm.
Period: Overall Study
Arm/Group | Boostrix I Group | Boostrix II Group
Started | 75 | 7
Completed | 73 | 7
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Boostrix I Group | Boostrix II Group | Total
Number analyzed (Participants) | 75 | 7 | 82
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.1 (0.31) | 21.1 (0.38) | 21.1 (0.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 6 | 72
  Male | 9 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-diphtheria (Anti-DT) and Anti-tetanus Toxoids (Anti-TT) Antibody Concentrations Above the Cut-offs
Description: The antibody concentrations cut-offs assessed were: equal to or above (≥) 0.1 international units per milliliter (IU/mL) and ≥ 1 IU/mL.
Time Frame: At Month 0
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity, which included all evaluable subjects who had received the booster dose of Boostrix™ vaccine and for whom immunogenicity data were available.
Measure: Number; unit: Subjects
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 74 | 7
Subjects
  Anti-diphtheria ≥ 0.1 IU/mL | 61 | 5
  Anti-diphtheria ≥ 1 IU/mL | 17 | 0
  Anti-tetanus ≥ 0.1 IU/mL | 72 | 7
  Anti-tetanus ≥ 1 IU/mL | 44 | 4

2. Primary Outcome: Number of Subjects With Anti-diphtheria (Anti-DT) and Anti-tetanus Toxoids (Anti-TT) Antibody Concentrations Above the Cut-offs
Description: as for outcome 1
Time Frame: At Month 1
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 73 | 7
Subjects
  Anti-diphtheria ≥ 0.1 IU/mL | 73 | 7
  Anti-diphtheria ≥ 1 IU/mL | 68 | 7
  Anti-tetanus ≥ 0.1 IU/mL | 73 | 7
  Anti-tetanus ≥ 1 IU/mL | 71 | 7

3. Secondary Outcome: Anti-diphtheria (Anti-DT) and Anti-tetanus Toxoids (Anti-TT) Antibody Concentrations
Description: Concentrations are presented as international units per millilitre (IU/mL).
Time Frame: At Month 0 (PRE) and Month 1 (POST)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 74 | 7
IU/mL
  Anti-diphtheria Pre [N=74;7] | 0.318 [0.24 to 0.421] | 0.196 [0.068 to 0.568]
  Anti-diphtheria Post [N=73;7] | 5.994 [4.679 to 7.68] | 3.226 [1.741 to 5.975]
  Anti-tetanus Pre [N=74;7] | 1.246 [0.956 to 1.623] | 0.989 [0.498 to 1.961]
  Anti-tetanus Post [N=73;7] | 9.596 [7.986 to 11.531] | 8.975 [5.277 to 15.264]

4. Secondary Outcome: Number of Seropositive Subjects for Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN)
Description: A seropositive subject was defined as a subject with anti-PT, anti-FHA and anti-PRN antibody concentrations ≥ 5 ELISA unit per milli-liter (EL.U/ml)
Time Frame: At Month 0 (PRE) and Month 1 (POST)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 75 | 7
Subjects
  Anti-PT Pre [N=75;7] | 46 | 7
  Anti-PT Post [N=73;7] | 73 | 7
  Anti-FHA Pre [N=75;7] | 75 | 7
  Anti-FHA Post [N=73;7] | 73 | 7
  Anti-PRN Pre [N=75;7] | 72 | 7
  Anti-PRN Post [N=73;7] | 73 | 7

5. Secondary Outcome: Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per millilitre (EL.U/mL).
Time Frame: At Month 0 (PRE) and Month 1 (POST)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 75 | 7
EL.U/mL
  Anti-PT Pre [N=75;7] | 9.1 [6.9 to 11.9] | 12.5 [8.8 to 17.9]
  Anti-PT Post [N=73;7] | 90.3 [73.9 to 110.5] | 116.5 [56.5 to 240.5]
  Anti-FHA Pre [N=75;7] | 63.8 [53.1 to 76.8] | 118.8 [80.6 to 175.1]
  Anti-FHA Post [N=73;7] | 793.4 [670.3 to 939.2] | 584.3 [248.3 to 1374.9]
  Anti-PRN Pre [N=75;7] | 36.9 [27.7 to 49.2] | 41.8 [20.3 to 85.9]
  Anti-PRN Post [N=73;7] | 548.1 [456.9 to 657.5] | 685.3 [243.5 to 1928.4]

6. Secondary Outcome: Number of Subjects With Booster Response to Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN)
Description: Booster response was defined as appearance of antibodies in subjects who were seronegative at the pre-vaccination time point (i.e. with concentrations < 5 El.U/mL) or at least 2-fold increase of prevaccination antibody concentrations in subjects who were seropositive at the pre-vaccination time point (i.e. with concentrations ≥5 El.U/mL.
Time Frame: At Month 1
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 73 | 7
Subjects
  Anti-PT [N=73;7] | 72 | 7
  Anti-FHA [N=73;7] | 71 | 6
  Anti-PRN [N=73;7] | 68 | 7

7. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 4-day (Day 0-3) follow-up period after booster vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects for whom data were available and with the symptom sheet filled in.
Measure: Number; unit: Subjects
Groups:
- Boostrix Pooled Group: Boostrix I and Boostrix II Groups pooled together.
Arm/Group | Boostrix Pooled Group
Number analyzed (Participants) | 81
Subjects
  Any pain | 76
  Grade 3 pain | 8
  Any redness | 48
  Grade 3 redness | 14
  Any swelling | 46
  Grade 3 swelling | 15

8. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], headache and gastrointestinal symptoms. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Day 0-3) follow-up period after booster vaccination
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Boostrix Pooled Group
Number analyzed (Participants) | 81
Subjects
  Any Fatigue | 44
  Grade 3 Fatigue | 2
  Related Fatigue | 36
  Any Fever | 7
  Grade 3 Fever | 0
  Related Fever | 7
  Any Gastrointestinal symptoms | 14
  Grade 3 Gastrointestinal symptoms | 1
  Related Gastrointestinal symptoms | 8
  Any Headache | 27
  Grade 3 Headache | 0
  Related Headache | 22

9. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 31-day (Day 0-30) follow-up period after booster vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Boostrix Pooled Group
Number analyzed (Participants) | 82
Subjects | 26

10. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: For safety assessment Boostrix I Group and Boostrix II Group were pooled (Pooled Group)
Population: as for outcome 9
Measure: Number; unit: Subjects
Arm/Group | Boostrix Pooled Group
Number analyzed (Participants) | 82
Subjects | 1

ADVERSE EVENTS:
Time Frame: Solicited local/general symtopms: during the 4-day post vaccination period. Unsolicited AE(s): during the 31-day post vaccination period. SAEs: during the entire study period (from Month 0 to Month 1).
Arm/Group | Boostrix Pooled Group
Serious Adverse Events (participants affected / at risk) | 1/82
Other Adverse Events (participants affected / at risk) | 78/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Boostrix Pooled Group (N=82)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Boostrix Pooled Group (N=82)
Pain (General disorders) | 76
Redness (General disorders) | 48
Swelling (General disorders) | 46
Fatigue (General disorders) | 44
Fever (Axillary) (General disorders) | 7
Gastrointestinal symptoms (General disorders) | 14
Headache (General disorders) | 27
Influenza (Infections and infestations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.